CLINICAL TRIAL: NCT02963597
Title: Auto-PAP for Pulmonary Hypertension Treatment in Decompensated Heart Failure Patients With Obstructive Sleep Apnea: A Two Center Pilot Study
Brief Title: Auto-PAP for Pulmonary Hypertension Treatment in Decompensated HF Patients With Sleep Apnea.
Acronym: ASAP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Resmed Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4889
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea, Obstructive; Hypertension, Pulmonary; Heart Failure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Intervention Model Description: CPAP Device
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Standard medical therapy plus AirSense™ 10 AutoSet for 48hrs.
  Interventions: Device: AirSense™ 10 AutoSet; Other: Standard Medical Therapy
- Group B (Placebo Comparator): Standard medical therapy only.
  Interventions: Other: Standard Medical Therapy

INTERVENTIONS:
Device: AirSense™ 10 AutoSet — The AirSense 10 AutoSet is a device that provide non-invasive ventilatory support to treat patients with sleep disordered breathing. The device is intended for home and hospital use. The treatment pressure required by the patient may vary due to changes in sleep state, body position and airway resistance. In AutoSet mode, the device provides only that amount of pressure required to maintain upper airway patency. The AirSense 10 AutoSet provides a minimum and maximum pressure within the range of 4-20 cm of water.
  Arms: Group A
Other: Standard Medical Therapy — Standard medical therapy according to current guidelines.

SUMMARY:
The objective of the study is to evaluate the effect of continuous positive airway pressure (PAP) therapy on pulmonary arterial (PA) pressures in acute decompensated heart failure (HF) patients with obstructive sleep apnea (OSA). The study will also assess changes in functional parameters, biomarkers, and echocardiographic parameters.

DETAILED DESCRIPTION:
The ASAP-HF study is a prospective, randomized, controlled, two-center, study with a parallel group design, with subjects randomized to either control (no APAP) or active treatment (APAP) in a 1:1 ratio. Group A (active): standard medical therapy plus treatment with continuous APAP for 48hrs, or Group B (control): standard medical therapy only.

Many people who have heart failure (HF) also have sleep-disordered breathing (SDB), which is breathing irregularities during sleep. These irregularities may interrupt the sleep as well as increase the rate of progression of Heart Failure. The ASAP-HF study is being done to see if certain clinical outcomes are improved in acute decompensated heart failure (HF) patients with SDB by using a non-invasive breathing device continuously for a short period of time (48 hours) while patient is still in the hospital. The device is called AirSense™ 10 AutoSet (AutoSet). It consists of an air flow generator, air tubing, an air humidifier, and a mask. As the patient breathe through the mask, the AutoSet monitors breathing.

The primary objective of this pilot study is to evaluate the effect of continuous positive airway pressure (PAP) therapy on pulmonary arterial (PA) pressures in acute decompensated heart failure (HF) patients with obstructive sleep apnea (OSA). The study will also assess changes in functional parameters, biomarkers, and echocardiographic parameters . This device is not currently used to diagnose sleep apnea and its utility is not well studied. This study will establish the utility of the device in diagnosing sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more
2. Decompensated Congestive Heart Failure with systolic Pulmonary Artery pressures of ≥50 mmHg (including Right Atrial pressure)
3. Prior clinical diagnosis of heart failure
4. Moderate to Severe predominately obstructive sleep disordered breathing documented by polygraphy with Apnea Hypopnea Index (AHI) ≥20e/h and 5% of the time spent <90% O2 Sat (minimum 2hr recording time)
5. Patient is able to fully understand study information and sign informed consent

Exclusion Criteria:

1. Chronic renal insufficiency (Hemodialysis or serum creatinine > 2)
2. Hemodynamically significant valvular disease
3. Severe arthritis or inability to complete 6 Minute Walk Test
4. Left Ventricular Assist Device/ heart transplant or hemodynamically unstable
5. Patient taking any Pulmonary vasodilators, including home oxygen.
6. Known diagnosis of Obstructive Sleep Apnea (OSA) and on active therapy
7. 80% of the respiratory events being central/Cheyne-Stokes breathing
8. Recent cardiac surgery (within 30 days of admission)
9. Recent stroke (within 30 days of admission or with persistent neurological deficits)
10. Severe Chronic Obstructive Pulmonary Disease defined as forced expiratory volume at one second (FEV1) < 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (2):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States
- Heart and Diabetes Center NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma S, Fox H, Aguilar F, Mukhtar U, Willes L, Bozorgnia B, Bitter T, Oldenburg O. Auto positive airway pressure therapy reduces pulmonary pressures in adults admitted for acute heart failure with pulmonary hypertension and obstructive sleep apnea. The ASAP-HF Pilot Trial. Sleep. 2019 Jul 8;42(7):zsz100. doi: 10.1093/sleep/zsz100. PMID 31004141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the inpatient clinical services of the Albert Einstein Medical Center Philadelphia (US) and from the Heart and Diabetes Center of North Rhine-Westphalia (Germany). Patients signed an informed consent for the study prior to any study-related procedure. Before randomization, all eligibility criteria were confirmed.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Standard medical therapy plus AirSense™ 10 AutoSet for 48hrs.
  AirSense™ 10 AutoSet: The AirSense 10 AutoSet is a device that provides non-invasive ventilatory support to treat patients with sleep-disordered breathing. The device is intended for home and hospital use. The treatment pressure required by the patient may vary due to changes in the sleep state, body position and airway resistance. In AutoSet mode, the device provides only that amount of pressure required to maintain upper airway patency. The AirSense 10 AutoSet provides a minimum and maximum pressure within the range of 4-20 cm of water.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (11.5) | 64.9 (9.96) | 67.75 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
  Germany | 5 | 6 | 11
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] — defined by weight (kg) / [height x height (m)]
  kg/m2 | 28.7 (5.8) | 31.2 (4.2) | 30.0 (5.0)
Type of heart failure according to EF (HFrEF/HFpEF) [Count of Participants; unit: Participants] — Heart failure with preserved ejection fraction/HFpEF (ejection fraction more than 45%).
  Heart failure with reduced ejection fraction/HFrEF (ejection fraction less than 45%)
  Participants
    HFpEF | 5 | 3 | 8
    HFrEF | 5 | 8 | 13
Smoking history [Count of Participants; unit: Participants]
  Active smoker | 1 | 2 | 3
  Former smoker | 3 | 3 | 6
  Never smoker | 6 | 6 | 12
History of COPD [Count of Participants; unit: Participants]
  Diagnosis of COPD confirmed with PFTs | 4 | 1 | 5
  No diagnosis of COPD or negative PFTs | 6 | 10 | 16
Apnea-hypopnea index (AHI) [Mean (Standard Deviation); unit: events/hour] — Apnea-hypopnea index (AHI) obtained by polygraphy (ApneaLink Air device).
  events/hour | 31.7 (8) | 34.3 (9.2) | 33.1 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Artery Systolic Pressure.
Description: The primary objective of this pilot study is to evaluate the effect of continuous positive airway pressure (PAP) therapy on pulmonary arterial (PA) pressures in acute decompensated heart failure (HF) patients with severe obstructive sleep apnea (OSA). The study will also assess changes in functional parameters, biomarkers, and echocardiographic parameters.
Time Frame: 48 hours
Population: Patients pulmonary artery systolic pressures were measured by transthoracic echocardiography (TTE) on admission and 48 hours after enrollment.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
mmHg
  Baseline | 58.6 [53.6 to 63.5] | 62.7 [56.2 to 69.2]
  After 48 hours | 42.8 [37.4 to 48.1] | 57.5 [49.9 to 65.1]

2. Secondary Outcome: Functional Parameters (6 Minute Walk Test) From Baseline to 48hrs
Description: 6-minute walk tests were performed on admission and repeated after 48 hours from the initial. The walked distance was measured in meters.
Time Frame: 48 hours
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
meters
  Baseline | 202.6 [151.5 to 253.6] | 153.6 [96.3 to 210.9]
  After 48 hours | 222.6 [156.9 to 288.2] | 161.8 [104.5 to 219.1]

3. Secondary Outcome: N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) From Baseline to 48hrs
Description: To compare changes in N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) measured at baseline and compared to 48hrs after.
Time Frame: 48 hours
Measure: Mean (95% Confidence Interval); unit: picogram/mililiter
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
picogram/mililiter
  Baseline | 1087.6 [528.29 to 1646.9] | 1532.7 [735.5 to 2329.9]
  After 48 hours | 466.5 [258 to 675] | 1500.2 [274.1 to 2726.2]

4. Secondary Outcome: Length of Stay
Description: The total stay in the hospital during the admission will be measured by days.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
days | 9.2 [5.3 to 13] | 13.7 [2.2 to 25.2]

5. Secondary Outcome: Blood Oxygenation.
Description: Changes in arterial blood oxygenation will be compared via arterial blood gas analysis performed at baseline and after 48h to assess arterial pressure of oxygen.
Time Frame: 48 hours
Population: Data was not available for all participants.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
mmHg
  Baseline: number analyzed (Participants) | 5 | 6
  Baseline | 72.84 [59.5 to 86.1] | 76.7 [69.9 to 83.5]
  After 48 hours: number analyzed (Participants) | 5 | 6
  After 48 hours | 80 [64.5 to 95.5] | 77.9 [71.2 to 84.5]

6. Secondary Outcome: Heart Failure Symptoms
Description: Heart failure symptoms as assessed by the New York Heart Association scale (NYHA) classification at baseline and after 48 hours. NYHA scale ranges from Class I to IV. Higher classes are associated with worst outcomes.
  Class I: No symptoms and no limitation in ordinary physical activity. Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity.Comfortable only at rest.
  Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: 48 hours
Population: Data was not available for participants after 48 hours. PI has left the institution; efforts to contact unsuccessful; data information not available for after 48hr time point
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
units on a scale
  Baseline | 3.2 [2.9 to 3.4] | 3.5 [3.2 to 3.8]
  After 48 hours: number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Fluid Retention
Description: Change in fluid retention as measured by weight at baseline and after 48 hours.
Time Frame: 48 hours
Population: Data after 48 hours was not available for the participants of the study. PI has left the institution; efforts to contact unsuccessful; data information not available for after 48hr time point
Measure: Mean (95% Confidence Interval); unit: Kg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
Kg
  Baseline | 82.6 [70.3 to 94.9] | 94.7 [81.6 to 107.8]
  After 48 hours: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: E/e' as an Assumption of LVEDP.
Description: Measurement of E/e' in 2D echocardiography as an assumption of LVEDP and PV acceleration time comparing baseline and after 48hrs.
Time Frame: 48 hours
Population: Data was not available for all the subjects at baseline and 48 hours after. PI has left the institution; efforts to contact unsuccessful; clarifying data information not available
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 11
Ratio
  Baseline: number analyzed (Participants) | 9 | 10
  Baseline | 18.6 [14.5 to 22.5] | 18.2 [13.6 to 22.7]
  After 48 hours: number analyzed (Participants) | 5 | 8
  After 48 hours | 14.8 [11.2 to 18.3] | 16.5 [13.9 to 19.0]

9. Post Hoc Outcome: Ejection Fraction in HFrEF
Description: Calculated ejection fraction in patients with heart failure with reduced ejection fraction (<45%) at baseline and after 48 hours.
Time Frame: 48 hours
Population: Analyzing only patients with heart failure with reduced ejection fraction (<45%).
Measure: Mean (95% Confidence Interval); unit: percentage (%)
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
percentage (%)
  Baseline: number analyzed (Participants) | 5 | 8
  Baseline | 23 [17.12 to 28.88] | 26.8 [18.4 to 35.3]
  After 48 hours: number analyzed (Participants) | 5 | 8
  After 48 hours | 30 [26.6 to 32.9] | 26.7 [18.3 to 35.2]

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
PI has left the institution; efforts to contact unsuccessful; additional data information not available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT02963597/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT02963597/SAP_001.pdf